CLINICAL TRIAL: NCT00004361
Title: Study of the Relationship Between Calcium Levels and Intact Parathyroid Hormone (iPTH) in Adults With Repaired or Palliated Conotruncal Cardiac Defects
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/11936; NU-553
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-01

CONDITIONS: Hypoparathyroidism; Tetralogy of Fallot; Pulmonary Valve Stenosis; Conotruncal Cardiac Defects; Heart Defects, Congenital; Pulmonary Atresia
Keywords: DiGeorge syndrome; cardiovascular and respiratory diseases; conotruncal cardiac defects; endocrine disorders; genetic diseases and dysmorphic syndromes; hypoparathyroidism; pulmonary valve stenosis; rare disease; tetralogy of Fallot
MeSH Terms: conditions — Hypoparathyroidism; Tetralogy of Fallot; Pulmonary Valve Stenosis; Conotruncal cardiac defects; Heart Defects, Congenital; Pulmonary Atresia; DiGeorge Syndrome; Respiratory Tract Diseases; Endocrine System Diseases; Genetic Diseases, Inborn; Rare Diseases | interventions — Calcium Gluconate; Sodium Citrate

INTERVENTIONS:
Drug: calcium gluconate
Drug: sodium citrate

SUMMARY:
OBJECTIVES: I. Identify latent hypoparathyroidism in normocalcemic adult survivors with repaired conotruncal cardiac defects, by evaluating parathyroid gland secretory function after induced hypocalcemia.

II. Determine the relationship of parathyroid hormone secretion to microdeletions in the same region of chromosome 22q11 as found in patients with DiGeorge anomaly.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients are given sodium citrate over a 2 hour infusion on day 1. Blood is drawn at times -30, -15, 0, and every 10 minutes thereafter during the infusion. On day 2, patients are given calcium gluconate over a 2 hour infusion. Blood is drawn at times -30, -15, 0, and every 10 minutes thereafter during the infusion.

ELIGIBILITY:
* Diagnostically shown repaired or palliated conotruncal cardiac defects, including tetralogy of Fallot with pulmonary stenosis or pulmonary atresia, truncus arteriosus, or interrupted aortic arch type B

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 1995-07

CONTACTS AND LOCATIONS:
Overall Officials: Craig B. Langman, Study Chair — Ann & Robert H Lurie Children's Hospital of Chicago